CLINICAL TRIAL: NCT06331910
Title: Topical Insulin in Treatment of Neurotrophic Corneal Ulcer,Efficacy And Safety
Brief Title: Efficacy and Safety of Topical Insulin for Neurotrophic Corneal Ulcers
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Abd Elrahim Ahmed, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TITNCUES
Record Dates: First submitted 2024-03-15; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Neurotrophic Keratopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- insulin eye drop (Experimental)
  Interventions: Drug: insulin eye drops

INTERVENTIONS:
Drug: insulin eye drops — Insulin eye drops deliver insulin directly to the cornea, They exploit insulin's ability to stimulate cell growth, potentially reducing healing time with minimal side effects.

SUMMARY:
To evaluate Safety and efficacy of topical insulin in treatment of neurotrophic corneal ulcers

DETAILED DESCRIPTION:
Neurotrophic keratopathy is a degenerative disease of the corneal epithelium resulting from impaired corneal innervation. A reduction In corneal sensitivity or complete corneal anesthesia is the hallmark of this disease and is responsible for producing epithelial keratopathy, ulceration and perforation.

Because decreased corneal sensitivity is the hallmark sign of neurotrophic keratitis (NK), corneal sensitivity testing should be performed as soon as It is suspected

There are 2 common ways to test-one qualitative, the other quantitative:

The qualitative method is most commonly used In clinic and often achieved with a cotton tipped applicator because It is easily accessible.

The most common quantitative method is the handheld esthesiometer (Cochet-Bonnet).

Standard treatment of neurotrophic corneal ulcer involves aggressive lubrication of the corneal surface, therapeutic contact lenses, amniotic membrane grafts and tarsorrhaphy . Refractory neurotrophic corneal ulcers occur when treatment response is incomplete and are potentially blinding.

Insulin is a widely available, relatively safe, and familiar medication that has been shown to improve corneal epithelial healing In vitro and in diabetic animal models. However, clinical experience with topical insulin in patients with non-healing corneal wounds is minimal.

Insulin-like growth factor-1 (IGF-1) has been shown to be an important modulator of corneal wound healing.

Topical insulin may be a simple and effective treatment for neurotrophic corneal ulcers.

The main outcome measurements for improvement are the decrease of ulcer size by fluroscien stain,the increase in visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurotrophic corneal ulcers caused by:

  * Herpes simplex or Herpes zoster viral infection
  * Topical anesthetics abuse
  * Chemical and physical burn
  * Chronic CL wear
  * Following LASIK,PRK,CXL
  * Following vitrectomy and endophotocoagulation for retinal detachment
  * Diabetes mellitus
  * Leprosy
  * Trigeminal neuralgia surgery

Exclusion Criteria:

* Non compliant patients with the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in ulcer size and the increase in visual acuity . | baseline
  To evaluate the effect of topical insulin eye drops in treatment of neurotrophic corneal ulcer.

REFERENCES:
- [Background] Wang AL, Weinlander E, Metcalf BM, Barney NP, Gamm DM, Nehls SM, Struck MC. Use of Topical Insulin to Treat Refractory Neurotrophic Corneal Ulcers. Cornea. 2017 Nov;36(11):1426-1428. doi: 10.1097/ICO.0000000000001297. PMID 28742619
- [Background] Shanley LJ, McCaig CD, Forrester JV, Zhao M. Insulin, not leptin, promotes in vitro cell migration to heal monolayer wounds in human corneal epithelium. Invest Ophthalmol Vis Sci. 2004 Apr;45(4):1088-94. doi: 10.1167/iovs.03-1064. PMID 15037573
- [Background] Zagon IS, Klocek MS, Sassani JW, McLaughlin PJ. Use of topical insulin to normalize corneal epithelial healing in diabetes mellitus. Arch Ophthalmol. 2007 Aug;125(8):1082-8. doi: 10.1001/archopht.125.8.1082. PMID 17698755
- [Background] Nishida T, Yanai R. Advances in treatment for neurotrophic keratopathy. Curr Opin Ophthalmol. 2009 Jul;20(4):276-81. doi: 10.1097/icu.0b013e32832b758f. PMID 19537364